CLINICAL TRIAL: NCT05725876
Title: Quantitative Fluorescence Molecular Imaging of Ustekinumab-800CW to Elucidate the Drug Distribution Throughout Inflamed Tissue in Crohn's Disease and Psoriasis: a Prospective Pilot Intervention Study
Brief Title: Quantitative Fluorescence Molecular Imaging of Ustekinumab-800CW to Elucidate the Drug Distribution Throughout Inflamed Tissue in Crohn's Disease and Psoriasis.
Acronym: VIDEO
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 83371
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Psoriasis; Crohn Disease
MeSH Terms: conditions — Psoriasis; Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Intervention Model Description: 15 naive patients before treatment and 10 patients on treatment in both diseases. Next to this we will also include 3 control patients in each disease. So 28 procedures for each disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Crohn's disease eligible for ustekinumab therapy (Experimental)
  Interventions: Drug: Ustekinumab
- Patients with Psoriasis eligible for Ustekunimab treatment (Experimental)
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Patients not on therapy and patients on therapy will undergo fluorescence molecular imaging.

SUMMARY:
Crohn's Disease (CD) and psoriasis are chronic inflammatory diseases. Ustekinumab is a humanized monoclonal antibody. Ustekinumab is expensive and primary non-response is high in both CD and psoriasis. Currently, there are no predictors of response to ustekinumab and the actual mechanism of action has not yet been elucidated. To clarify the mechanism of action and gain a better understanding of the high primary non-response rates, the University Medical Center Groningen (UMCG) developed a tracer fluorescently labeling ustekinumab. This study aims to gain insight into ustekinumab distribution and concentrations in the gut. The current study aims to identify the ustekinumab target cells in the inflamed gut mucosa and skin using quantitative fluorescence molecular endoscopy (qFME). By gaining insight into local ustekinumab concentrations, drug distribution, and by discovering target cells, we expect to gain insight into the mechanism of action of ustekinumab.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of CD or PsO
* Non-responsive to conventional therapy
* Active disease:

  * CD cohort: clinically active disease of the bowel defined either clinically as at least moderate activity using dedicated scoring indices (for definitions of disease activity, see below) or biochemically active disease as defined by a faecal calprotectin > 200 ug/g;
  * PsO: clinically active disease of at least PASI ≥ 10 or clinically active disease as assessed by a dermatologist;
* Age ≥ 18 years;
* Written informed consent.

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent according to treating medical physician;
* Prior ustekinumab treatment within the last 15 weeks (except for patients in the treatment arm and control group);
* Ustekinumab contraindicated as therapy;
* Pregnancy or breast feeding. A negative pregnancy test must be available for women of childbearing potential (i.e. premenopausal women with intact reproductive organs and women less than two years after menopause);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-06 (Estimated)

PRIMARY OUTCOMES:
Quantification of fluorescent signal of fluorescent ustekinumab in CD and psoriasis patients. | 3-4 days after tracer admission

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No